CLINICAL TRIAL: NCT03397069
Title: Efficacy of Midazolam Addition to Local Anesthetic in Peribulbar Block. Randomized, Controlled Trial
Brief Title: Midazolam Additive to Local Anesthetic in Peribulbar Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al Jedaani Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AlJedaaniH
Record Dates: First submitted 2017-12-23; First posted 2018-01-11 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-01

CONDITIONS: Postoperative Pain; Cataract; Local Anaesthetic Complication; Midazolam
Keywords: peribubar block - midazolam
MeSH Terms: conditions — Pain, Postoperative; Cataract | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group C(control) (Placebo Comparator): Peribulbar block without midazolam (peribulbar block using a mixture of lidocaine 2%, hyaluronidase 15 IU / ml)
  Interventions: Procedure: Peribulbar block (control)
- Group M1 (Experimental): Peribulbar block with midazolam 50 µg (peribulbar block using a mixture of lidocaine 2%, hyaluronidase 15 IU / ml. plus midazolam 50 µg/ml)
  Interventions: Procedure: Peribulbar block(M1)
- Group M2 (Experimental): Peribulbar block with midazolam 100 µg(peribulbar block using a mixture of lidocaine 2%, hyaluronidase 15 IU / ml. plus midazolam 100 µg/ml
  Interventions: Procedure: Peribulbar block(M2)

INTERVENTIONS:
Procedure: Peribulbar block (control) — The Peribulbar block was performed by inserting the needle percutaneously at the area bounded by 1- The imaginary perpendicular line joining inferior lacrimal papilla to the inferior margin of the orbit, laterally 2- Lateral border of the nose, medially 3- Inferior lacrimal canaliculus, superiorly and 4- Inferior orbital margin, inferiorly. The needle was introduced in an anteroposterior direction to its half-length and then in an oblique direction to the optical foramen.
  After negative aspiration, 6-8 ml of local anesthetic solution (lidocaine 2%, hyaluronidase 15 IU / ml ) was injected slowly over about 40 seconds or until the appearance of lid fullness. This was followed by a gentle digital massage to the eyeball to facilitate diffusion of the local anesthetic mixture.
  Other Names: Peribulbar block without midazolam
  Arms: Group C(control)
Procedure: Peribulbar block(M1) — The Peribulbar block was performed by inserting the needle percutaneously at the area bounded by 1- The imaginary perpendicular line joining inferior lacrimal papilla to the inferior margin of the orbit, laterally 2- Lateral border of the nose, medially 3- Inferior lacrimal canaliculus, superiorly and 4- Inferior orbital margin, inferiorly. The needle was introduced in an anteroposterior direction to its half-length and then in an oblique direction to the optical foramen.
  After negative aspiration, 6-8 ml of local anesthetic solution (lidocaine 2%, hyaluronidase 15 IU / ml. plus midazolam 50 µg/ml ) was injected slowly over about 40 seconds or until the appearance of lid fullness. This was followed by a gentle digital massage to the eyeball to facilitate diffusion of the local anesthetic mixture.
  Other Names: Peribulbar block with midazolam 50ug
  Arms: Group M1
Procedure: Peribulbar block(M2) — The Peribulbar block was performed by inserting the needle percutaneously at the area bounded by 1- The imaginary perpendicular line joining inferior lacrimal papilla to the inferior margin of the orbit, laterally 2- Lateral border of the nose, medially 3- Inferior lacrimal canaliculus, superiorly and 4- Inferior orbital margin, inferiorly. The needle was introduced in an anteroposterior direction to its half-length and then in an oblique direction to the optical foramen.
  After negative aspiration, 6-8 ml of local anesthetic solution (lidocaine 2%, hyaluronidase 15 IU / ml. plus midazolam 100 µg/ml ) was injected slowly over about 40 seconds or until the appearance of lid fullness. This was followed by a gentle digital massage to the eyeball to facilitate diffusion of the local anesthetic mixture.
  Other Names: Peribulbar block with midazolam 100ug
  Arms: Group M2

SUMMARY:
Regional eye blocks are usually preferred for ophthalmic procedures. Peribulbar block (PBB) is a safe alternative for patients undergoing cataract surgery. Many studies tried to solve this issue by means of prolonging the duration of action of the local anesthetics used. Several drugs were tried as adjuncts to local anesthetics, and their effects have been studied. Midazolam added to the list of adjuvant used in the subarachnoid or epidural block can produce analgesia, probably mediated by the benzodiazepine-Gamma Amino-Butyric Acid(GABA) receptor complex.

The investigators hypothesized that the addition of midazolam to lidocaine will improve the quality of the peribulbar block; fasten the onset and prolonging its anesthetic and analgesic duration.

ELIGIBILITY:
Inclusion Criteria:

* 90 adult patients with ASA physical status I to III
* Aged 40-70 years
* Scheduled for elective extracapsular or phacoemulsification cataract surgery with peribulbar block
* No history of allergy to local anesthetics
* Axial length less than 28 mm.

Exclusion Criteria:

* Patient's refusal to share in the study
* communication barrier (e.g. impaired hearing, disturbed conscious level, impaired mental status)
* uncontrolled tremors
* morbidly obese patients
* allergy to lidocaine
* coagulation abnormalities
* glaucoma
* recent surgical procedure on the same eye.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Quality of the sensory and motor block | 6 hours
  The quality of the sensory and motor block was assessed using the Ocular Anesthesia Scoring System (OASS). Patients were categorized into three groups according to the quality of the block and level of anesthesia achieved: poor (0-3), average (4-9) and good block (10-14)

SECONDARY OUTCOMES:
Onset and duration of block | 6 hours
  The onset of motor block (globe akinesia), sensory block, and lid akinesia (ptosis). Were recorded from the time of injection of (LAS) until complete globe akinesia, a disappearance of sensation, and complete lid akinesia (ptosis). Duration of globe akinesia was recorded till recurrence of muscle movements (score 8). Similarly, the return of sensation to the globe was assessed by digital spear pressure at the limbus.
Analgesia | 4 hours postoperative
  Postoperative pain was assessed at 30 minutes' intervals utilizing verbal rating scale (VAS) on a scale of 0 to 10 (where 0 means no pain and 10 means the worst imaginable pain) for a period of 4 hours postoperative or until first analgesic request
local or systemic complications | 6 hours
  sub-conjunctival hematoma, itching, ecchymosis, diplopia, blindness, nausea, vomiting, dry mouth, and hypotension, were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Al Jedaani group of hospitals, Jeddah, Meccah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ibrahim M, Gomaa E. Efficacy of midazolam addition to local anesthetic in peribulbar block : Randomized controlled trial. Anaesthesist. 2019 Mar;68(3):143-151. doi: 10.1007/s00101-018-0525-3. Epub 2019 Jan 9. PMID 30627737